CLINICAL TRIAL: NCT00689767
Title: COronary Native Artery First in Man Investigation of ISA 247 Elution to Prevent Restenotic Mechanisms
Brief Title: COronary Native Artery First in Man Investigation of ISA 247 Elution to Prevent Restenotic Mechanisms (CONFIRM 1)
Acronym: CONFIRM 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated ahead of schedule after completion of the 3-year follow-up time point due to Sponsor decision.
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 801; Application #: 2008-001347-20
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): This arm will receive the coated stent
  Interventions: Device: CINATRA™ ISA 247 Coated Coronary Stent System
- B (Active Comparator): This arm will receive a bare metal stent
  Interventions: Device: CINATRA™ Coronary Stent System

INTERVENTIONS:
Device: CINATRA™ Coronary Stent System — Bare metal cobalt chromium stent implantation
  Arms: B
Device: CINATRA™ ISA 247 Coated Coronary Stent System — Drug coated cobalt chromium stent implantation
  Arms: A

SUMMARY:
This First In Man study is a prospective, multicentre, single blind, randomized, controlled clinical trial of the CINATRA™ ISA 247 Coated Coronary Stent System as compared to the CINATRA™ Coronary Stent System. The study will enroll up to 100 evaluable patients at up to 7 sites. Clinical follow up will occur at 1 month, 6 months, and 1, 2, 3, 4 and 5 years post procedure. Repeat angiography and IVUS will be performed at the 6 month follow up time point for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable angina pectoris (Canadian Cardiovascular Society 1, 2, 3) or unstable angina pectoris with documented ischemia (CCS 4, Braunwald Class IB-C, IIB-C or IIIB-C), or patients with documented silent ischemia.
2. Patients who are eligible for coronary revascularization (percutanous angioplasty).
3. Acceptable candidates for coronary artery bypass grafting (CABG).
4. Patients with de novo lesion in a native coronary artery >50% and <100% stenosis.

   NOTE: Treatment of lesions in a non-target vessel is up to the investigator's discretion (max. two-vessel-disease).

   ONLY a bare metal stent (no drug eluting stent) can be used for this treatment. Treatment of any non-target vessel lesions must be successfully completed before enrolling patient and placing study stent.
5. The target lesion must be a maximum length of 13 mm (visual estimate) and able to be covered by one stent.
6. The reference diameter of the target lesion must be 3.0 mm by visual estimate.
7. Left ventricular ejection fraction of >30%.
8. Patients willing to provide written informed consent prior to participation and willing and able to participate in all follow-up evaluations.

Exclusion Criteria:

1. Patients under the age of 18 or unable to give informed consent.
2. Women who are pregnant. Women of child bearing potential must have a negative pregnancy test within 7 days prior to enrollment and utilize reliable contraception at a minimum until after the angiographic follow up.
3. Patients who previously participated in this study.
4. Patient is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints.

   NOTE: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.
5. Life expectancy of less than 12 months or factors making clinical and/or angiographic follow-up difficult (no fixed address, etc.).
6. Patients who intend to have a major surgical intervention within 6 months of enrollment in the study.
7. Patients with new ST elevation within 48 hours prior to stenting.
8. Braunwald Class IA, IIA and IIIA angina pectoris.
9. Patients with a contraindication to an emergency coronary bypass surgery.
10. Patients who had previous Coronary Artery Bypass Surgery (CABG).
11. Any individual who may refuse a blood transfusion.
12. Serum creatinine >3.0 mg/dL.
13. Platelet count <100,000 cells/mm³.
14. Patients with intolerance or contraindication to acetylsalicylic acid (aspirin), heparin, cyclosporin or cyclosporine derivative, clopidogrel or ticlopidine drug therapy.
15. Patients with contrast agent hypersensitivity that cannot be adequately pre-medicated.
16. Patients who have a stent anywhere within the target vessel.
17. Any planned interventional treatment of any vessel post study procedure.

    Exclusion Criteria Related to Angiography
18. Patients with previous PCI of the same segment (i.e. no restenotic lesions).
19. Previous interventional procedure (less than 6 months) anywhere within the target vessel;
20. Target lesion is located in or supplied by an arterial or venous bypass graft.
21. Target lesion involves a side branch >2.0mm in diameter.
22. Ostial target lesion (within 3.0mm of vessel origin).
23. Target vessel has evidence of thrombus or is excessively tortuous that makes it unsuitable for proper stent delivery and deployment .
24. Patients with total occlusions (TIMI 0).
25. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off.
26. Target lesion requires treatment with a device other than the predilatation balloon prior to stent placement (including but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, cutting balloon etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Van Langenhove, MD, Principal Investigator — Middelheim Hospital, Antwerp, Belgium
Locations (7):
- Belgium (7):
  - Middelheim Hospital, Antwerp
  - Imelda ziekenhuis, Bonheiden
  - Cliniques universitaires Saint-Luc, Brussels
  - Ziekenhuis Oost Limburg, Campus Sint Jan, Genk
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Virga Jesse Ziekenhuis, Hasselt
  - UZ Leuven Cardiovascular Institute, Leuven